CLINICAL TRIAL: NCT01669759
Title: The Study in the Correlation Between the Severity of Post-stroke Fatigue and the Severity of qi Deficiency and Blood Stasis in Chinese Medicine.
Brief Title: The Study in the Correlation Between the Severity of Post-stroke Fatigue and the Severity of qi Deficiency and Blood Stasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DMR101-IRB2-151
Record Dates: First submitted 2012-08-14; First posted 2012-08-21 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Poststroke Fatigue

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- fatigue

SUMMARY:
The purpose of the present study was to investigate the correlation between the severity of fatigue, and the severity of qi deficiency and blood stasis.

DETAILED DESCRIPTION:
According to the reports of department of Health, stroke has been the top three ranking in leading ten major mortality causes. Although fatigue is a common symptom after stroke, but it is easy to neglect due to fatigue is a non-specific symptom. Based on the literature review, fatigue symptom is not only common on post-stroke patient and it also has highly correlation with mortality, prognosis and efficacy of rehabilitation. In Traditional Chinese Medicine recording, Wang Qing-ren suggests that the main etiology of stroke is results from qi stagnation and blood stasis, thereafter, the study about qi deficiency and blood stasis became to the main stream for stroke until now. Therefore, the purpose of the present study was to investigate the correlation between the severity of fatigue, and the severity of qi deficiency and blood stasis.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: men or women
2. Age:40~80 years old
3. Stroke history at least 3 months
4. Hemorrhage or ischemic stoke
5. Conscious clear and can communicate
6. Brief Fatigue Inventory-Taiwan form score ≥ 4
7. Sign informed consent

Exclusion Criteria:

1. Patient with psychotic diagnosis and can't cooperate with researcher
2. Major disease: chronic obstructive pulmonary disease, heart failure, myocardial infarction, chronic renal failure, liver cirrhosis
3. Pregnant women
4. Breastfeeding women

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with post-stroke fatigue were enrolled from the departments of neurological, neurosurgical, and rehabilitation in China Medical University Hospital (Taichung, Taiwan), their Brief Fatigue Inventory-Taiwan form score ≥ 4, and stroke onset more than 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Frome Fatigue severity level scale to evaluate fatigue severity score. | about 20 minutes
  When patient visit first time,we complete all the evaluation scale. Total evaluation time is about 20 minutes. And all data will be analyzed one year later.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan, Taiwan